CLINICAL TRIAL: NCT05925348
Title: Effect of Endotoxinemia on the Incidence of Postoperative Vasoplegia or Vasoplegic Shock Following Cardiothoracic Surgery Using Cardiopulmonary Bypass
Brief Title: Endotoxinemia and Vasoplegia Following Cardiothoracic Surgery With Cardiopulmonary Bypass (CPB)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Other Study IDs: AnIt22-11
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Vasoplegia; Vasoplegic Shock
Keywords: Endotoxin; cardiopulmonary bypass (CBP); Vasoplegia; Vasoplegic shock
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with cardiopulmonary bypass — Due to the observational design of the study, no study-specific interventions are performed.
  Blood samples are measured to analyze blood-levels of endotoxin

SUMMARY:
This observational study investigates the effect of endotoxinemia on the postoperative incidence of vasoplegia or vasoplegic shock in patients undergoing cardiac surgery with the use of cardiopulmonary bypass.

DETAILED DESCRIPTION:
Through previous research, it has been well established that cardiothoracic surgery using cardiopulmonary bypass (CPB) causes a systemic inflammatory response. This is in part due to the surgical trauma, the extracorporeal circulation and factors that come with it (e.g. blood contact with foreign surfaces, mechanical stress etc.), and ischemia. This inflammatory response is a key contributor to the incidence of vasoplegia and vasoplegic shock following these types of surgery - a common complication that in turn causes significant morbidity and mortality. Over the years, many factors that contribute to this reaction have been discussed. One potential explanation is the release of endotoxin into the bloodstream during CPB. Endotoxin is a molecule that is a part of bacteria which are native to the human gut. In healthy subjects, cell-barriers prevent release of relevant amounts of endotoxin into the blood stream. During major interventions, and especially during cardiac surgery with CPB, this barrier function is impeded, allowing endotoxin levels to rise and potentially exert detrimental effects. While previous studies have indicated that endotoxin may in fact be released into the bloodstream in significant concentrations, and there are some mechanistic explanations to how endotoxin may contribute to the resulting inflammation and vasoplegia, available studies have been small and the evidence is inconclusive. This study aims to show whether different blood-levels of endotoxin are associated with vasoplegia and vasoplegic shock in patients undergoing cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients undergoing cardiac surgery requiring CPB
2. written informed consent

Exclusion Criteria:

1. emergency surgery in the context of acute coronary syndrome
2. patients with chronic inflammatory diseases of the gut
3. patients receiving immunosuppressive drugs
4. patients with infectious endocarditis
5. patients with sepsis
6. patients with chronic kidney disease with estimated glomerular filtration rate (eGFR) <20 ml/min/1,73m²
7. persons with any kind of dependency on the investigator or employed by the institution responsible or investigator
8. persons held in an institution by legal of official order -

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Perioperative patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Norepinephrine equivalent dose (NED) | within 24 hours following induction of general anesthesia

SECONDARY OUTCOMES:
Fluid input | within 24 hours following induction of general anesthesia
Fluid balance | within 24 hours following induction of general anesthesia
Occurence of Acute Kidney Injury (AKI) according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria | 72 hours after cardiac surgery
Duration of mechanical ventilation | within 72 hours after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Therapy and Pain Medicine
Locations (1):
- University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No